CLINICAL TRIAL: NCT02774174
Title: Post Marketing Clinical Follow Up for the Evaluation of the METS™ Proximal Humeral System Using Retrospective Data
Brief Title: The Evaluation of the METS™ Proximal Humeral System
Status: Completed | Type: Observational
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-02
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Complications; Arthroplasty
Keywords: Proximal Humerus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- METS Proximal Humeral system: Implanted with METS Proximal Humerus

SUMMARY:
This study is a single centre, non-randomised, post market clinical follow up examining retrospective patient data from a series of surgical cases; which involved the endoprosthetic replacement of the proximal humerus using the Stanmore Implant Worldwide METS (Modular Endoprosthetic Tumour System) Proximal Humeral system.

The objective of this study is to evaluate the retrospective patient data where patients have been followed up for at least 12 months post operation; to demonstrate the safety of the METS Proximal Humeral replacement system.

DETAILED DESCRIPTION:
The METS™ Proximal Humeral system is an endoprosthetic replacement designed to restore the length and the function of an arm after the resection of a significant amount of bone tissue; due to a malignant tumour in the proximal humerus. This Post Market Clinical Follow up (PMCF) study is designed to further support the existing evidence that the system is safe and performs as expected, when analysing retrospective patient data that have had a METS™ Proximal Humeral replacement. The target population is male or female subjects aged between 18 years and over who have been implanted with a METS™ Proximal Humeral system at the Royal National Orthopaedic Hospital, Stanmore; and the patient has been followed up for at least 12 months following implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 and over who has been implanted with a METS™ Proximal Humeral system implant at the Royal National Orthopaedic Hospital, Stanmore.
2. Patient has been followed up for at least 12 months following implant surgery
3. Patient had their surgery on or after January 2007

Exclusion Criteria:

1. Patient is currently or has been involved in pending litigation or worker's compensation
2. Patient has participated in another clinical investigation or study with an investigational medical device within the last 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects aged between 18 years and over who have been implanted with a METS™ Proximal Humeral system at the Royal National Orthopaedic Hospital, Stanmore; and the patient has been followed up for at least 12 months following implantation
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation of adverse events that occurred within 12 months post implantation | Follow Up of 12 months
  Adverse events within the first 12 months will be assessed and evaluated

CONTACTS AND LOCATIONS:
Overall Officials: William JS Aston, MBBSMRCSFRCS, Principal Investigator — Royal National Orthopaedic Hospital
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a retrospective safety evaluation study. Data will already be deidentified before the clinical research team receive it.